CLINICAL TRIAL: NCT01256918
Title: Evaluation of Phacodepth Required to Achieve Full Thickness Nuclear Crack in Various Grades of Cataract and to Determine the Correlation Between the Two.
Brief Title: Study of Phacodepth Required for Safe and Effective Chop During Phacoemulsification for Cataract.
Acronym: CALIBCHOP
Status: Completed | Type: Observational
Sponsor: Dr. Ram Manohar Lohia Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Praveen Kumar Malik, Professor and Consultant,ophthalmology, Dr. Ram Manohar Lohia Hospital
Other Study IDs: RMLH-001-EYE
Record Dates: First submitted 2010-12-07; First posted 2010-12-09 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-07

CONDITIONS: Cataract
Keywords: cataract; phacoemulsification; phacochop; phacotip
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There is a correlation between phacodepth required for full thickness nuclear crack and the various grades of cataract

DETAILED DESCRIPTION:
BACKGROUND:- Phacochop techniques have been categorized as either horizontal or vertical. These approaches are thought to be among the best techniques for managing hard cataracts. In vertical chop technique proper placement of the phaco tip is crucial. It must be embedded deeply into the centre of the nucleus , pointing toward the optic nerve , with high vacuum and burst mode.Inadequate penetration of phacotip may result in partial thickness nuclear crack with residual posterior plate and overzealous penetration may result in posterior capsular rupture.This may be avoided if some estimate can be made preoperatively of the depth of penetration required to achieve full thickness crack. With this in mind the study intends to make a preoperative assessment of the depth required to reach the centre of the nuclei and observe the actual depth of penetration required for a safe and effective vertical chop.

MATHEMATICAL BASIS :- The cross section of a lens nucleus is ellipsoidal . A geometrical estimate of the radius of the ellipse (x )traversed by the phacotip to reach the centre can be made preoperatively.The calculation would depend largely on three parameters.

The major axis of the ellipse ( namely the lens diameter[b] ) The minor axis of the ellipse (namely lens thickness[a] ) The point of entry on the surface of the lens.This defines an angle Ø which this radius makes with the vertical axis and in turn can be approximated by the length of the arc from centre of lens surface to entry point[y].

Adult human crystalline lens varies in thickness from 4.2+/-0.5 mm and has a diameter of 9.6+/- 0.4mm. Assuming the lens diameter (b) to be from 9.2 mm to 10.0mm , the lens thickness ( a) varying from 3.7mm to 4.7mm and the point of entry of phacotip 2.0mm to 3.0mm from centre of anterior lens surface ( y ) , this distance (x) would vary from 2.59mm to 3.2mm.(using Online Wolfram calculator) in thinnest to thickest nuclei. This would be increased with increase in ( a ) as well as ( y ) .In cataractous lens the harder a nucleus the deeper it may be required to penetrate to achieve a full thickness crack.

If the investigators make a note of all three variables i.e lens thickness , nuclear hardness and point of entry at the time of surgery and correlate with the actual depth required at the time of surgery the investigators may be able to recommend an effective and safe phacodepth for achieving full thickness nuclear crack in various grades of hard cataract.

Till now it was not possible to measure the length of penetration of phacotip during surgery. The investigators have designed a calibrated phacotip with visible markings on 0.2mm scale from 2 to 3. 4mm to enable measurements and recordings.

Thus the investigators aim to identify a safe and effective phacodepth required in each grade of cataract {3.0 - 6.9 according to Lens Opacities Classification System( LOCS-III )}to achieve successful nuclear crack . At the same time any correlation between different nuclear grades and the effective phacodepth would be analysed to find any association between them.

ELIGIBILITY:
Inclusion Criteria:

* Patients (> 40 years of age) with grade 3.0 to 6.9( according to LOCS-III) of senile cataract will be included in this study

Exclusion Criteria:

1. Subluxated and dislocated lens.
2. Central leukomatous corneal opacity preventing visualization of cataractous lens for grading and surgery.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at EYE DEPARTMENT, Post Graduate Institute of Medical Education and Research(PGIMER) , Dr R.M.L Hospital.
  A consecutive sample of all eyes with cataract reporting to the eye OPD of Dr. R.M.L.Hospital and fulfilling the inclusion criteria, would be enrolled in the study starting a date following ethics committee approval till March 2011 ,after a written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Praveen K Malik, MS, Principal Investigator — Dr. R.M.L.Hospital,New Delhi,India
Locations (1):
- Dr. R.M.L.Hospital,, New Delhi, National Capital Territory of Delhi, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A consecutive sample of 200 eyes with cataract reporting to the eye outpatient department (OPD) of Dr. Ram Manohar Lohia (R.M.L.)Hospital and fulfilling the inclusion criteria, were enrolled in the study starting Nov.2010 till January 2011 ,after a written informed consent.
Groups:
- Patients Undergoing Phacoemulsification: Patients (> 40 years of age) with grade 3.0 to 6.9( according to LOCS-III) of senile cataract were included in this study.200 consecutive patients were enrolled and achievement of milestone noted while attempting vertical chop during phacoemulsification using a calibrated phacotip.
Period: Overall Study
Arm/Group | Patients Undergoing Phacoemulsification
Started | 200
Full Thickness Nuclear Crack Achieved | 200
Completed | 200
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Undergoing Phacoemulsification
Number analyzed (Participants) | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 113
  >=65 years | 87
Age Continuous [Mean (Standard Deviation); unit: years] | 62.7 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 89
Region of Enrollment [Number; unit: participants]
  India | 200

OUTCOME MEASURES:

1. Primary Outcome: Phacodepth Required to Achieve Full Thickness Nuclear Crack
Description: phacodepth is the term used to describe the depth penetrated by the phacotip into the substance of lens.A note of depth penetrated by the tip to achieve full thickness nuclear crack shall be made.
Time Frame: day 0 of surgery
Population: A consecutive sample of all eyes with cataract reporting to the eye OPD of Dr. R.M.L.Hospital and fulfilling the inclusion criteria, were enrolled in the study starting Nov.2010 till Jan 2011 ,after a written informed consent.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Phacodepth: A note shall be made of the phacodepth at which a complete vertical chop is achieved during the attempted vertical chop .
Arm/Group | Phacodepth
Number analyzed (Participants) | 200
mm | 2.5755 (0.1816)

2. Secondary Outcome: Posterior Capsular Rupture
Description: A note shall be made of any posterior capsular rupture attributable to the attempted vertical chop .
Time Frame: day 0 of surgery.
Population: . In this observational study sample size was achieved by consecutive sampling of all eyes with cataract reporting to the eye OPD of Dr. R.M.L.Hospital and fulfilling the inclusion criteria from Nov.2010 till March 2011 ,after a written informed consent.
  Occurence of any posterior capsular rupture during vertical chop was noted as per protocol.
Measure: Number; unit: participants
Groups:
- Posterior Capsular Rupture: A note shall be made of any posterior capsular rupture attributable to the attempted vertical chop during the phacoemulsification procedure.
Arm/Group | Posterior Capsular Rupture
Number analyzed (Participants) | 200
participants | 0
Statistical Analysis 1: Comparison: Posterior Capsular Rupture; Any occurence of posterior capsular rupture in attempted vertical chop would have been an indicator of overzealous penetration as the vertical chop even though effective would not have been safe. We hypothesised that use of callibrated phacotip after careful preoperative assessment for performing vertical chop during phacoemulsification is not associated with any posterior capsular rupture we noted any incidence of posterior capsular rupture; Test type: Superiority or Other; p > 0.05, incidence; incidence = 0

3. Primary Outcome: Correlation Between Nuclear Colour and Phacodepth Required for a Safe and Effective Vertical Chop During Phacoemulsification
Description: the nuclear colour grading as per LOCS III criteria for each case and the depth of penetration of phacotip required during a vertical chop was analysed to look for any correlation between the two.
Time Frame: day 0 of surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Nuclear Colour: nuclear grading as per LOCS III criteria for cataract shall be done on a decimal scale from 0.1 to 6.9 nuclear colour is graded on a scale from 0.1 to 6.9 by comparing with standard photographs of cataract, under lens opacities classification system III, on a Haag Streit slit lamp under standard conditions of illumination
- Phacodepth: actual depth of penetration(in mm) of phacotip required to achieve a full thickness crack in vertical chop during phacoemulsification
Arm/Group | Nuclear Colour | Phacodepth
Number analyzed (Participants) | 200 | 200
units on a scale | 4.7565 (1.2225) | 2.5755 (0.1816)
Statistical Analysis 1: Comparison: Nuclear Colour vs Phacodepth; null hypothesis : there is no correlation between nuclear colour and phacodepth required for a full thickness crack during a vertical chop; Test type: Superiority or Other; p < 0.05, pearson correlation coefficient; pearson correlation coefficient = 0.850958

4. Primary Outcome: Correlation Between Nuclear Opalescence and Phacodepth
Description: Pearson correlation coefficient would be calculated to look for any correlation between
  1. nuclear opalescence as per LOCS III grading system for each cataract and
  2. penetration of phacotip required to achieve a full thickness nuclear crack in vertical chop during phacoemulsification of the cataractous lens
Time Frame: day 0 of surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Nuclear Opalescence: nuclear grading as per LOCS III criteria for cataract.nuclear opalescence is graded on a scale from 0.1 to 6.9 by comparing with standard photographs of cataract, under lens opacities classification system III, on a Haag Streit slit lamp under standard conditions of illumination
- Phacodepth: actual depth of penetration (in mm) of phacotip required to achieve a full thickness crack in vertical chop during phacoemulsification
Arm/Group | Nuclear Opalescence | Phacodepth
Number analyzed (Participants) | 200 | 200
units on a scale | 4.665 (1.2150) | 2.5755 (0.1816)
Statistical Analysis 1: Comparison: Nuclear Opalescence vs Phacodepth; Null hypothesis: there is no correlation between nuclear opalescence and phacodepth required to achieve full thickness nuclear crack using a callibrated phacotip; Test type: Superiority or Other; p < 0.05, pearson correlation coefficient; pearson correlation coefficient = 0.842617

5. Primary Outcome: Correlation Between Lens Thickness and Phacodepth
Description: Pearson correlation coefficient would be calculated to look for any correlation between
  1. length thickness measurement using A scan biometer for each cataract and
  2. penetration of phacotip required to achieve a full thickness nuclear crack in vertical chop during phacoemulsification of the cataractous lens
Time Frame: day 0 of surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lens Thickness: lens thickness as measured using an A scan biometer
- Phacodepth: depth of penetration of phacotip required to achieve a full thickness crack in vertical chop during phacoemulsification
Arm/Group | Lens Thickness | Phacodepth
Number analyzed (Participants) | 200 | 200
units on a scale | 3.9799 (0.5082) | 2.5755 (0.1816)
Statistical Analysis 1: Comparison: Lens Thickness vs Phacodepth; null hypothesis there is no correlation between lens thickness and penetration of phacotip (phacodepth)required to achieve full thickness crack in vertical chop during phacoemulsification; Test type: Superiority or Other; p > 0.05, pearson correlation coefficient; pearson correlation coefficient = 0.111166

ADVERSE EVENTS:
Time Frame: any occurrence of corneal epithelial damage due to A scan biometry during preoperative assessment was noted during the period from day of examination to 24hrs. thereafter for each participant during the entire period of recruitment.
Arm/Group | Patients Undergoing Phacoemulsification
Serious Adverse Events (participants affected / at risk) | 0/200
Other Adverse Events (participants affected / at risk) | 0/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Undergoing Phacoemulsification (N=200)
posterior capsular rupture (Eye disorders) | 0 (0)

LIMITATIONS AND CAVEATS:
first time use of callibrated phacotip to measure phacotip penetration during vertical chop during phacoemulsification , hence no pre existing results to compare with.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes